CLINICAL TRIAL: NCT04042922
Title: Acute Treatment of Alzheimer's Disease With Gamma Frequency Stimulation
Brief Title: High Frequency Light and Sound Stimulation to Improve Brain Functions in Alzheimer's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1902706647
Record Dates: First submitted 2019-07-24; First posted 2019-08-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Cognitive Impairment; Non-invasive Sensory Stimulation; Light and Sound Stimulation; Gamma
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Exposure to active stimulation for 30 - 60 min (Experimental): Subjects in this arm will receive 30 - 60 minutes of active stimulation
  Interventions: Device: GENUS device (Active Settings)
- Exposure to control stimulation for 30 - 60 min (Sham Comparator): Subjects in this arm will receive 30 - 60 minutes of control stimulation
  Interventions: Device: GENUS device (Sham Settings)

INTERVENTIONS:
Device: GENUS device (Active Settings) — Participants in the experimental group will use the GENUS device configured to active settings for 30 - 60 minutes.
  Other Names: Gamma frequency stimulation; Light and sound stimulation
  Arms: Exposure to active stimulation for 30 - 60 min
Device: GENUS device (Sham Settings) — Participants in the control group will use the GENUS device configured to sham settings for 30 - 60 minutes.
  Other Names: Gamma frequency stimulation; Light and sound stimulation
  Arms: Exposure to control stimulation for 30 - 60 min

SUMMARY:
Alzheimer's disease (AD) is characterized by significant memory loss and toxic protein deposits (amyloid and tau) in the brain. The investigators' lab found a non-invasive way to remove these toxic proteins from the brain in AD mouse models. Remarkably, treated mice also have improved memory on behavioral testing. The investigators aim to translate this non-invasive method, which uses light and sound to stimulate the brain, to be used in mild Alzheimer's patients. 40 participants with mild Alzheimer's disease will be recruited, and the investigators will assess their brain waves with electroencephalogram (EEG) before, during, and after light and sound stimulation for safety, feasibility, and to optimize the stimulation device for use in the mild AD population.

DETAILED DESCRIPTION:
It is known that Alzheimer's disease (AD) patients have significant disruptions in brain waves, especially the gamma frequency (~30 - 100 Hz) waves. Recently, the investigators' lab found that gamma entrainment using light and sound stimulation, which the investigators call GENUS, improves memory and decreases toxic accumulation of amyloid and tau in AD mouse models. This study aims to translate these findings in the mouse models to be used in mild Alzheimer's patients. The investigators will recruit 40 patients diagnosed with mild AD who will be randomly assigned to two study arms. Cognitive and mental health evaluations as well as memory tests will be performed on all subjects. All subjects will also be exposed to the GENUS device, which can deliver light and sound waves at different frequencies. The GENUS device is composed of a panel with light-emitting diode (LED) illumination and speakers for auditory stimulation. Each of the 2 groups will have different combinations of light and sound settings. The investigators will use electroencephalography (EEG) to check for how the participant's brain waves respond to the stimulation, and use questionnaires to evaluate for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 50 - 100.
* Subject must have mild Alzheimer's disease with a Mini Mental State Exam (MMSE) score of 19 -26.
* Subject is willing to sign informed consent document.
* If subject is deemed to not have capacity to sign the informed consent, he/she will need a legally authorized representative to provide surrogate consent.

Exclusion Criteria:

* Subjects who do not have healthcare.
* Subjects who are being treated with N-methyl-D-aspartate (NMDA) receptor antagonists (eg. Memantine).
* Subjects on medications that lower seizure threshold such as wellbutrin, ciprofloxacin, levofloxacin, etc.
* Subjects with history of seizure or epilepsy within the past 24 months.
* Subjects with clinically significant suicide risk and/or suicide attempt in the past 1 year.
* Subjects with behavioral problems such as aggression/agitation/impulsivity that might interfere with their ability to comply with protocol.
* Active treatment with one or more anti-epileptic agent.
* Subjects who have had a stroke within the past 24 months.
* Subjects diagnosed with migraine headache.
* Active treatment with one or more psychiatric agent (e.g. antidepressants, antipsychotics, etc).
* Subjects who have an active implantable medical device including but not limited to implantable cardioverter defibrillator (ICD), deep brain stimulator (DBS), cardiac pacemaker, and/or sacral nerve stimulator.
* Subjects who have profound hearing or visual impairment.
* Subjects who have a life expectancy of less than 2 years.
* Subjects who are pregnant.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of gamma frequency stimulation | Immediately after the completion of the stimulation
  Feasibility of gamma frequency stimulation in subjects with mild AD will be assessed by analyzing the EEG data from each subject for a sign of change in gamma frequency waves and determining the percent of subjects who show this change.
Tolerability of gamma frequency stimulation | Immediately after the completion of the stimulation
  Tolerability of gamma frequency stimulation will be assessed by using a questionnaire asking for the subjects' overall experience with the stimulation.
Safety of gamma frequency stimulation | Immediately after the completion of the stimulation
  Safety of gamma frequency stimulation will be assessed by using a questionnaire asking for any adverse effects of the stimulation.

OTHER OUTCOMES:
Changes in working memory after gamma frequency stimulation | Baseline and immediately after the completion of the stimulation
  Exploratory measure to check if there is any change in n-back test performance, between baseline and immediately after the completion of the stimulation.
  The n-back test involves a sequence of stimuli (e.g., letters, numbers), presented one at a time, and a subject is asked to indicate when the current stimulus is the same as the stimulus presented n times earlier in the sequence. The performance metrics will include the "hit" rate (number of correct responses out of total number of target stimuli; ranging from 0 to 1), "false alarm" rate (number of incorrect responses out of total number of non-target stimuli; ranging from 0 to 1), and response time.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Huei Tsai, PhD, Principal Investigator — Massachusetts Institute of Technology; Edward S Boyden, PhD, Principal Investigator — Massachusetts Institute of Technology; Diane Chan, MD, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Derived] Chan D, Suk HJ, Jackson BL, Milman NP, Stark D, Klerman EB, Kitchener E, Fernandez Avalos VS, de Weck G, Banerjee A, Beach SD, Blanchard J, Stearns C, Boes AD, Uitermarkt B, Gander P, Howard M 3rd, Sternberg EJ, Nieto-Castanon A, Anteraper S, Whitfield-Gabrieli S, Brown EN, Boyden ES, Dickerson BC, Tsai LH. Gamma frequency sensory stimulation in mild probable Alzheimer's dementia patients: Results of feasibility and pilot studies. PLoS One. 2022 Dec 1;17(12):e0278412. doi: 10.1371/journal.pone.0278412. eCollection 2022. PMID 36454969